CLINICAL TRIAL: NCT03266276
Title: Assessing the Impact of Cancer Care Ontario's Psychosocial Oncology & Palliative Care Pathway in Ambulatory Head and Neck Cancer Clinics
Brief Title: Assessing Impact of CCO's PSO & PC Pathway in Ambulatory HNC Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 267-2016
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Cancer; Supportive Care
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
  After completing HNC staff interprofessional team training in PSO and PC, an RCT will be used to examine the impact of using a standardized PSOPC pathway approach, prompted follow up with patients and documentation. Participants will be recruited and randomized into (1) care as usual group and (2) "intervention" PSOPC pathway group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual Control Group (No Intervention): Treatment as usual.
- Intervention Group (Experimental): Use of a standardized PSOPC pathway approach, prompted follow up with patients and documentation.
  Interventions: Other: PSOPC pathway approach

INTERVENTIONS:
Other: PSOPC pathway approach — The intervention will use a standardized PSOPC pathway approach, prompted follow up with patients and documentation.
  Additionally, clinicians will be prompted to document conversations about response to emotional or physical ESAS symptom scores, symptom management plan (self/education/monitoring/medication), illness understanding; and, if necessary, an offer of PSO/PC referral.
  Arms: Intervention Group

SUMMARY:
Rates of depression and anxiety in cancer patients are much higher compared to the general population. 40% of head and neck cancer patients will develop significant distress along the cancer journey. Less than half of these patients are able to access support, with factors such as age, social difficulty, cancer stage and site affecting referral. In 2016, 78,000 Canadians died of cancer, yet there is limited implementation of routine and integrated advanced care planning in cancer care.

An upcoming deliverable of all cancer centres in Ontario is the integration of Cancer Care Ontario's Psychosocial and Palliative Care (PSOPC) pathway into all disease pathways. Successful widespread implementation of this pathway at Odette Cancer Centre (OCC) will impact >16,000 patients/year. If effective, it will reduce suffering, unnecessary healthcare utilization, improve treatment decisions and compliance, enable a better quality of life in survivorship and improve quality at end of life. There is a need for better developed, standardized response pathways to address PSO and PC needs throughout the patient's journey.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is the sixth most commonly diagnosed cancer worldwide. Individuals with HNC experience a high burden of symptom-related distress (e.g. emotional, physical, psychological, spiritual etc.). Additionally, HNC patients may experience facial disfigurement, communication barriers, social stigma, lack of social support, and/or self-imposed or experienced disease stigma. The presence of depression, anxiety or social difficulty is relatively common in HNC patients yet less than half of those with significant distress access psychosocial (PSO) and palliative care (PC). Few studies have examined a systematic response to reducing distress, integrating a routine psychosocial and palliative care approach to oncology, with planning for future care for this population.

Most cancer centres do not have a systematic model of practice geared towards distress screening, PC and PSO approach to care. Therefore, determining how to best incorporate PSO and PC (PSOPC) into the interprofessional oncology clinic management of patients with HNC remains an important and unanswered question. The question remains of how to proactively identify those at higher risk for distress and greater need for specialized psychosocial or palliative care. Some oncologists consider the provision of PSOPC as an integral part of their professional role. Yet increasing the delivery of quality primary PSOPC by busy oncologists may require targeted training, the use of algorithms to prompt PC and PSO assessment, incorporating response to distress screening / advanced care planning tools into routine clinical processes, prompts to document conversations about illness understanding and consideration of individual factors influencing treatment decisions.

The primary goal of this study is to integrate quality primary level PSO and PC into clinic care by developing and evaluating a routine response to screening in hopes of increasing documentation of the following: discussion of response to ESAS, illness understanding, advanced care planning or goals of care conversations.

Specifically, this study will examine the impact of Cancer Care Ontario's (CCO) PSOPC Pathway, an expert panel recommended algorithm for assessing and managing symptoms and initiating a PSOPC approach and timely specialized referral, when necessary.

Phase Two: Randomized Controlled Trial

After completing the needs assessment and interprofessional team training in PSO and PC, an RCT will be used to examine the impact of using a standardized PSOPC pathway approach, prompted follow up with patients and documentation. Participants will be recruited and randomized into care as usual group and "intervention" PSOPC pathway group.

Main Hypothesis:

It is hypothesized that compared to treatment as usual, the PSOPC pathway intervention group will result in an increase in (larger proportion of):

Rationale and Objective:

Innovation: Model of clinical service delivery Currently, there is no standardized process for meeting the psychosocial and palliative care needs of HNC. This project promotes learner,needs-driven professional development, and knowledge translation. It will foster a person-focused, results-driven, integrated and sustainable model of clinical service delivery.

Individual clinics and cancer centres have developed their own responses to Edmonton Symptom Assessment System (ESAS) distress screening. However, we believe this project is a unique Oncology Team/PC/PSO/Patient Advisor collaboration, where all members will work together to improve symptom assessment and management, improve discussions and documentation involving illness understanding and advanced care planning to better meet PSO and PC needs, whilst assessing the role for the PSOPC Pathway.

An additional innovation for this project is to develop and evaluate a customizable approach to assessing the needs of an oncology team, thereby shaping both professional development experiences and determining a model of care delivery that should be acceptable within the clinic frame.

Improving Healthcare and Patient Experience:

The CCO PSOPC pathway was designed to guide improvements in the provision of primary PSOPC Care, including symptom response, communication, illness understanding, advanced care planning, as well as increased identification of those who require access to specialized PSO and PC beyond the skill set of the oncology team. An inaccurate illness understanding (whether the cancer is curable or not and whether it is progressing) hinders informed discussions and decisions and supportive end of life planning. And, while some patients with moderate to severe ESAS ratings have their symptoms assessed and managed, this is not the case for all patients. Earlier advanced care planning discussions help patients and their families have a better understanding of the disease to make more personalized, informed decisions about care.

ELIGIBILITY:
Inclusion Criteria:

* Consenting ambulatory OCC HNC patients, with baseline ESAS scores of >2 (emotional) or >3 (physical symptoms) with no active suicidal ideation, cognitive impairment or significant debilitation such that participation would be burdensome for participants and/or safety concerns as determined by a research assistant.

Exclusion Criteria:

* If participants endorse thoughts of dying at baseline, they will be asked to complete semi-structured questions to assess suicidal ideation (SI). If there is any active SI or intent, the oncology team will be informed, a record kept and the participant will be withdrawn from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Increased documentation of response to symptoms (ESAS), PPS, illness understanding and advanced care planning (ACP) | baseline
  Documented high ESAS scores (>6) and of all PPS scores, symptom management and conversations about PSO-either distress/management/referral/resources, PC needs, and ACP, illness understanding

SECONDARY OUTCOMES:
The European Organization for Research and Treatment of Cancer Quality of Life (EORTC-QOL 30) | baseline, 1, 3, and 6 months
  Valid and reliable 30-item questionnaire assessing health related quality of life
  o 5 functional, 3 symptom, global HRQOL and single item scales
Princess Margaret Hospital Satisfaction with Doctor Questionnaire (PMH-PSQ 24) | baseline, 1, 3, and 6 months
  PMH-PSQ 24 taps domains of Interpersonal skills, time spent with physician, information and physician relationship likert-type response scale (strongly agree/agree/disagree/strongly disagree/does not apply) consisting of 24 items (49)
  o Measures two facets of satisfaction with care: physician disengagement and perceived support.
Mixed-methods interviews | 1 and 3 months
  Mixed-methods interview questions assess patients' perceptions of their overall treatment experience and care received at OCC
  * 10 open-ended questions assessing patients' perceptions of the compassion and empathy received from HCPs
  * 10 questions taken from CCO's Person-Centered Care and Patient Experience with Outpatient Cancer Care Index assessing three dimensions of care: communication, self-management and support for shared decision-making
  * 31 questions taken the Ambulatory Oncology Patient Satisfaction Survey (AOPSS) assessing patients' perceptions of emotional support; information, communication and education; respect for patient preferences; coordination and continuity of care; physical comfort and access to care
  * 3 questions from iLead Champions Conversations With Patients assessing whether patients felt their personal needs were heard and met by HCPs during treatment
Patient Health Questionnaire (PHQ-9) | baseline, 1, 3, and 6 months
  9 questions corresponding to the 9 diagnostic criteria for major depression DSMV as '0' (not at all) to '3' (nearly every day)
Beck Depression Inventory (BDI-II) | baseline, 1, 3, and 6 mnths
  If depression/anxiety ESAS 3 or above, BDI to further assess depressive symptoms and assess for change in scores
General Anxiety Disorder (GAD-7) | baseline, 1, 3, and 6 months
  To measure the severity of anxiety among patients 7-item tool based on DSM-V criteria has a scale similar to PHQ-9
Beck Anxiety Inventory (BAI) | baseline, 1, 3, and 6 months
  If depression/anxiety ESAS 3 or above, BAI to further assess anxiety symptoms and assess for change in scores
Experiences in Close Relationships Inventory | baseline, 1, 3, and 6 months
  Assessing how patients feel in close relationships with other people
Patient and, if participating, Caregiver Semi-structured interview | 1 and 3 months
  A series of qualitative and quantitative questions assessing patients' experiences during care and caregivers' perceptions of quality of care, illness understanding and whether patient psychosocial and palliative needs were met during treatment
Edmonton Symptom Assessment System | baseline, 1 and 3 months
  9 items designed to assess the severity of the most commonly reported symptoms experienced by cancer patients including pain, fatigue, drowsiness, nausea, dyspnea, depression, anxiety, well-being, and loss of appetite
Palliative Performance Scale | baseline
  Quantitatively represents a person's performance status and ability to function
  * 11 point scale from 100% (healthy) to 0% (death) with 10% decrements
  * The scale is based on five observable parameters: ambulation, ability to do activities, self-care, food/fluid intake, and consciousness level
Illness Understanding Questionnaire | 1, 3, and 6 months
  A series of questions assessing patients' understanding of the course, nature and treatment of their illness

CONTACTS AND LOCATIONS:
Overall Officials: Janet Ellis, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortholan C, Benezery K, Dassonville O, Poissonnet G, Bozec A, Guiochet N, Belkacemi Y. A specific approach for elderly patients with head and neck cancer. Anticancer Drugs. 2011 Aug;22(7):647-55. doi: 10.1097/CAD.0b013e328344282a. PMID 21394019
- [Background] Argiris A, Karamouzis MV, Raben D, Ferris RL. Head and neck cancer. Lancet. 2008 May 17;371(9625):1695-709. doi: 10.1016/S0140-6736(08)60728-X. PMID 18486742
- [Background] Devins GM, Payne AY, Lebel S, Mah K, Lee RN, Irish J, Wong J, Rodin GM. The burden of stress in head and neck cancer. Psychooncology. 2013 Mar;22(3):668-76. doi: 10.1002/pon.3050. Epub 2012 Mar 5. PMID 22392570
- [Background] Burlein-Hall, S. (January 2015). Unpublished data from Odette Cancer Centre symptom screening audit.
- [Background] Rhoten BA, Deng J, Dietrich MS, Murphy B, Ridner SH. Body image and depressive symptoms in patients with head and neck cancer: an important relationship. Support Care Cancer. 2014 Nov;22(11):3053-60. doi: 10.1007/s00520-014-2312-2. Epub 2014 Jun 14. PMID 24925049
- [Background] Lebel S, Castonguay M, Mackness G, Irish J, Bezjak A, Devins GM. The psychosocial impact of stigma in people with head and neck or lung cancer. Psychooncology. 2013 Jan;22(1):140-52. doi: 10.1002/pon.2063. Epub 2011 Sep 19. PMID 21932417
- [Background] Weiner B, Perry RP, Magnusson J. An attributional analysis of reactions to stigmas. J Pers Soc Psychol. 1988 Nov;55(5):738-48. doi: 10.1037//0022-3514.55.5.738. PMID 2974883
- [Background] Else-Quest NM, LoConte NK, Schiller JH, Hyde JS. Perceived stigma, self-blame, and adjustment among lung, breast and prostate cancer patients. Psychol Health. 2009 Oct;24(8):949-64. doi: 10.1080/08870440802074664. PMID 20205038
- [Background] Bultz BD, Waller A, Cullum J, Jones P, Halland J, Groff SL, Leckie C, Shirt L, Blanchard S, Lau H, Easaw J, Fassbender K, Carlson LE. Implementing routine screening for distress, the sixth vital sign, for patients with head and neck and neurologic cancers. J Natl Compr Canc Netw. 2013 Oct 1;11(10):1249-61. doi: 10.6004/jnccn.2013.0147. PMID 24142826
- [Background] Hammerlid E, Ahlner-Elmqvist M, Bjordal K, Biorklund A, Evensen J, Boysen M, Jannert M, Kaasa S, Sullivan M, Westin T. A prospective multicentre study in Sweden and Norway of mental distress and psychiatric morbidity in head and neck cancer patients. Br J Cancer. 1999 May;80(5-6):766-74. doi: 10.1038/sj.bjc.6690420. PMID 10360654
- [Background] Oishi A, Murtagh FE. The challenges of uncertainty and interprofessional collaboration in palliative care for non-cancer patients in the community: a systematic review of views from patients, carers and health-care professionals. Palliat Med. 2014 Oct;28(9):1081-98. doi: 10.1177/0269216314531999. Epub 2014 May 12. PMID 24821710
- [Background] Vigano A, Dorgan M, Buckingham J, Bruera E, Suarez-Almazor ME. Survival prediction in terminal cancer patients: a systematic review of the medical literature. Palliat Med. 2000 Sep;14(5):363-74. doi: 10.1191/026921600701536192. PMID 11064783
- [Background] Cancer Quality Council of Ontario. Access to Psychosocial Oncology Service (2016.) http://www.csqi.on.ca/by_patients_journey/diagnosis/acess_to_psychosocial_oncology_services/
- [Background] Dansky Ullmann C, Harlan LC, Shavers VL, Stevens JL. A population-based study of therapy and survival for patients with head and neck cancer treated in the community. Cancer. 2012 Sep 15;118(18):4452-61. doi: 10.1002/cncr.27419. Epub 2012 Jan 17. PMID 22252676
- [Background] Turnbull Macdonald GC, Baldassarre F, Brown P, Hatton-Bauer J, Li M, Green E, Lebel S. Psychosocial care for cancer: a framework to guide practice, and actionable recommendations for Ontario. Curr Oncol. 2012 Aug;19(4):209-16. doi: 10.3747/co.19.981. PMID 22876147
- [Background] Cancer Care Ontario (2013) Psychosocial Oncology & Palliative Care Pathway: Disease Pathway Management. https://www.cancercare.on.ca/ocs/qpi/dispathmgmt/disease_pathway_maps/psychosocial_palliative_pathway/
- [Background] Buchmann L, Conlee J, Hunt J, Agarwal J, White S. Psychosocial distress is prevalent in head and neck cancer patients. Laryngoscope. 2013 Jun;123(6):1424-9. doi: 10.1002/lary.23886. Epub 2013 Apr 1. PMID 23553220
- [Background] Carlson LE, Waller A, Groff SL, Bultz BD. Screening for distress, the sixth vital sign, in lung cancer patients: effects on pain, fatigue, and common problems--secondary outcomes of a randomized controlled trial. Psychooncology. 2013 Aug;22(8):1880-8. doi: 10.1002/pon.3223. Epub 2012 Nov 12. PMID 23147718
- [Background] Ellis J, Lin J, Walsh A, Lo C, Shepherd FA, Moore M, Li M, Gagliese L, Zimmermann C, Rodin G. Predictors of referral for specialized psychosocial oncology care in patients with metastatic cancer: the contributions of age, distress, and marital status. J Clin Oncol. 2009 Feb 10;27(5):699-705. doi: 10.1200/JCO.2007.15.4864. Epub 2008 Dec 29. PMID 19114706
- [Background] Canadian Cancer Society's Advisory Committee on Cancer Statistics. Canadian Cancer Statistics 2015. Toronto, On: Canadian Cancer Society;2015.
- [Background] Akechi T, Okuyama T, Sugawara Y, Nakano T, Shima Y, Uchitomi Y. Major depression, adjustment disorders, and post-traumatic stress disorder in terminally ill cancer patients: associated and predictive factors. J Clin Oncol. 2004 May 15;22(10):1957-65. doi: 10.1200/JCO.2004.08.149. PMID 15143090
- [Background] Kugaya A, Akechi T, Okuyama T, Nakano T, Mikami I, Okamura H, Uchitomi Y. Prevalence, predictive factors, and screening for psychologic distress in patients with newly diagnosed head and neck cancer. Cancer. 2000 Jun 15;88(12):2817-23. doi: 10.1002/1097-0142(20000615)88:123.0.co;2-n. PMID 10870066
- [Background] Derogatis LR, Morrow GR, Fetting J, Penman D, Piasetsky S, Schmale AM, Henrichs M, Carnicke CL Jr. The prevalence of psychiatric disorders among cancer patients. JAMA. 1983 Feb 11;249(6):751-7. doi: 10.1001/jama.249.6.751. PMID 6823028
- [Background] Zabora J, BrintzenhofeSzoc K, Curbow B, Hooker C, Piantadosi S. The prevalence of psychological distress by cancer site. Psychooncology. 2001 Jan-Feb;10(1):19-28. doi: 10.1002/1099-1611(200101/02)10:13.0.co;2-6. PMID 11180574
- [Background] Shim EJ, Shin YW, Jeon HJ, Hahm BJ. Distress and its correlates in Korean cancer patients: pilot use of the distress thermometer and the problem list. Psychooncology. 2008 Jun;17(6):548-55. doi: 10.1002/pon.1275. PMID 17957764
- [Background] Lam WW, Shing YT, Bonanno GA, Mancini AD, Fielding R. Distress trajectories at the first year diagnosis of breast cancer in relation to 6 years survivorship. Psychooncology. 2012 Jan;21(1):90-9. doi: 10.1002/pon.1876. Epub 2010 Dec 2. PMID 21132676
- [Background] Von Essen L, Larsson G, Oberg K, Sjoden PO. 'Satisfaction with care': associations with health-related quality of life and psychosocial function among Swedish patients with endocrine gastrointestinal tumours. Eur J Cancer Care (Engl). 2002 Jun;11(2):91-9. doi: 10.1046/j.1365-2354.2002.00293.x. PMID 12099944
- [Background] Onitilo AA, Nietert PJ, Egede LE. Effect of depression on all-cause mortality in adults with cancer and differential effects by cancer site. Gen Hosp Psychiatry. 2006 Sep-Oct;28(5):396-402. doi: 10.1016/j.genhosppsych.2006.05.006. PMID 16950374
- [Background] Faller H, Bulzebruck H, Drings P, Lang H. Coping, distress, and survival among patients with lung cancer. Arch Gen Psychiatry. 1999 Aug;56(8):756-62. doi: 10.1001/archpsyc.56.8.756. PMID 10435611
- [Background] Singer S, Krauss O, Keszte J, Siegl G, Papsdorf K, Severi E, Hauss J, Briest S, Dietz A, Brahler E, Kortmann RD. Predictors of emotional distress in patients with head and neck cancer. Head Neck. 2012 Feb;34(2):180-7. doi: 10.1002/hed.21702. Epub 2011 Mar 11. PMID 21400629
- [Background] Krebber AM, Jansen F, Cuijpers P, Leemans CR, Verdonck-de Leeuw IM. Screening for psychological distress in follow-up care to identify head and neck cancer patients with untreated distress. Support Care Cancer. 2016 Jun;24(6):2541-8. doi: 10.1007/s00520-015-3053-6. Epub 2015 Dec 23. PMID 26694718
- [Background] Merckaert I, Libert Y, Messin S, Milani M, Slachmuylder JL, Razavi D. Cancer patients' desire for psychological support: prevalence and implications for screening patients' psychological needs. Psychooncology. 2010 Feb;19(2):141-9. doi: 10.1002/pon.1568. PMID 19382112
- [Background] Junn JC, Kim IA, Zahurak ML, Tan M, Fan KY, Lake ST, Zaboli D, Messing BP, Ulmer K, Harrer KB, Gold D, Ryniak KL, Zinreich ES, Tang M, Levine MA, Blanco RG, Saunders JR, Califano JA, Ha PK. Multidisciplinary service utilization pattern by advanced head and neck cancer patients: a single institution study. Int J Otolaryngol. 2012;2012:628578. doi: 10.1155/2012/628578. Epub 2012 Oct 18. PMID 23118755
- [Background] Cancer Care Ontario (2009). A Quality Initiative of the Program in Evidence-Based care (PEBC), Cancer care Ontario (CCO): The Management of Head and Neck Cancer in Ontario. https://www.cancercare.on.ca/cmmon.pages/userfile.aspx?fileld=58592
- [Background] Cancer Quality Council of Ontario. Symptom Assessment and Management (2015). https://www.csqi.on.ca/by_patient_journey/treatment/symptom_assessment_and_managment/
- [Background] Madeline Li, manuscript in preparation
- [Background] Weeks JC, Cook EF, O'Day SJ, Peterson LM, Wenger N, Reding D, Harrell FE, Kussin P, Dawson NV, Connors AF Jr, Lynn J, Phillips RS. Relationship between cancer patients' predictions of prognosis and their treatment preferences. JAMA. 1998 Jun 3;279(21):1709-14. doi: 10.1001/jama.279.21.1709. PMID 9624023
- [Background] Myers J, Kim A, Flanagan J, Selby D. Palliative performance scale and survival among outpatients with advanced cancer. Support Care Cancer. 2015 Apr;23(4):913-8. doi: 10.1007/s00520-014-2440-8. Epub 2014 Sep 18. PMID 25228018
- [Background] Glare PA, Sinclair CT. Palliative medicine review: prognostication. J Palliat Med. 2008 Jan-Feb;11(1):84-103. doi: 10.1089/jpm.2008.9992. PMID 18370898
- [Background] Temel JS, Greer JA, Admane S, Gallagher ER, Jackson VA, Lynch TJ, Lennes IT, Dahlin CM, Pirl WF. Longitudinal perceptions of prognosis and goals of therapy in patients with metastatic non-small-cell lung cancer: results of a randomized study of early palliative care. J Clin Oncol. 2011 Jun 10;29(17):2319-26. doi: 10.1200/JCO.2010.32.4459. Epub 2011 May 9. PMID 21555700
- [Background] Cancer Care Ontario (2013) Palliative Care Collaborative Plans CCPS: Condensed Version. https:// www.cancercare.on.ca/common.pages/UserFile.aspx?fileld=57766
- [Background] Anderson F, Downing GM, Hill J, Casorso L, Lerch N. Palliative performance scale (PPS): a new tool. J Palliat Care. 1996 Spring;12(1):5-11. PMID 8857241
- [Background] Bainbridge D, Seow H, Sussman J, Pond G, Martelli-Reid L, Herbert C, Evans W. Multidisciplinary health care professionals' perceptions of the use and utility of a symptom assessment system for oncology patients. J Oncol Pract. 2011 Jan;7(1):19-23. doi: 10.1200/JOP.2010.000015. PMID 21532805
- [Background] Palliative Performance Scale (PPSv2). Medical Care of the Dying,4th ed.; p120. Copyright Victoria Hospice Society,2006. http://www.victoriahospice.org/ed_publications.html accessed November 25,2015
- [Background] Ripamonti CI, Bandieri E, Pessi MA, Maruelli A, Buonaccorso L, Miccinesi G. The Edmonton Symptom Assessment System (ESAS) as a screening tool for depression and anxiety in non-advanced patients with solid or haematological malignancies on cure or follow-up. Support Care Cancer. 2014 Mar;22(3):783-93. doi: 10.1007/s00520-013-2034-x. Epub 2013 Nov 26. PMID 24276952
- [Background] Abdollahzadeh F, Sadat Aghahossini S, Rahmani A, Asvadi Kermani I. Quality of life in cancer patients and its related factors. J Caring Sci. 2012 May 27;1(2):109-14. doi: 10.5681/jcs.2012.016. eCollection 2012 Jun. PMID 25276684
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Ruiz MA, Zamorano E, Garcia-Campayo J, Pardo A, Freire O, Rejas J. Validity of the GAD-7 scale as an outcome measure of disability in patients with generalized anxiety disorders in primary care. J Affect Disord. 2011 Feb;128(3):277-86. doi: 10.1016/j.jad.2010.07.010. Epub 2010 Aug 9. PMID 20692043
- [Background] Bitar R, Bezjak A, Mah K, Loblaw DA, Gotowiec AP, Devins GM. Does tumor status influence cancer patients' satisfaction with the doctor-patient interaction? Support Care Cancer. 2004 Jan;12(1):34-40. doi: 10.1007/s00520-003-0534-9. Epub 2003 Oct 30. PMID 14586667
- [Background] Haisfield-Wolfe ME, McGuire DB, Soeken K, Geiger-Brown J, De Forge BR. Prevalence and correlates of depression among patients with head and neck cancer: a systematic review of implications for research. Oncol Nurs Forum. 2009 May;36(3):E107-25. doi: 10.1188/09.ONF.E107-E125. PMID 19403439
- [Background] Epstein AS, Prigerson HG, O'Reilly EM, Maciejewski PK. Discussions of Life Expectancy and Changes in Illness Understanding in Patients With Advanced Cancer. J Clin Oncol. 2016 Jul 10;34(20):2398-403. doi: 10.1200/JCO.2015.63.6696. Epub 2016 May 23. PMID 27217454
- [Background] Krebber AM, Leemans CR, de Bree R, van Straten A, Smit F, Smit EF, Becker A, Eeckhout GM, Beekman AT, Cuijpers P, Verdonck-de Leeuw IM. Stepped care targeting psychological distress in head and neck and lung cancer patients: a randomized clinical trial. BMC Cancer. 2012 May 10;12:173. doi: 10.1186/1471-2407-12-173. PMID 22574757